CLINICAL TRIAL: NCT06813235
Title: Dream2Heal: A Pilot Sequential Multiple Assignment Randomized Trial (SMART) of an Adaptive Stepped-care Intervention for Chinese Cancer Survivors With Mild-to-moderate Insomnia
Brief Title: Dream2Heal: An Adaptive Stepped-care Intervention for Chinese Cancer Survivors With Mild-to-moderate Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 24-531
Record Dates: First submitted 2025-01-23; First posted 2025-02-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Neoplasm; Sleep Disturbance
Keywords: Sequential multiple assessment randomized controlled trial; sleep disturbance; cancer survivors; insomnia; Survivorship intervention
MeSH Terms: conditions — Neoplasms; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: First stage intervention: Participants will be randomised to either the iD2H (an unsupervised, self-guided web-based version of the D2H intervention based off cognitive behavioural therapy for insomnia (CBT-I)) or eEX intervention (an unsupervised, self-guided web-based exercise intervention), at a 1:1 ratio.
  Second stage intervention: Non-respondents to the initial intervention will be randomly assigned to either the D2H (face-to-face, therapist led CBT-I intervention) or augmented intervention (combined, unsupervised, self-guided web-based intervention that covers the content of iD2H and eEX interventions) as stepped-up care at a 1:1 ratio. Two sets of block randomisation sequences with randomly permuted block sizes of 2, 4 and 6 will be generated for both stages of the randomisation, where one set will be used for the first stage and the second set will be used for the second stage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, investigator and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to intervention or control arms.
  The participants are masked in terms of not knowing that one intervention is hypothesized to yield larger effects than the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First stage intervention: iDream2Heal (Experimental): iDream2Heal (iD2H) is an unsupervised, self-guided web-based intervention, consisting of five weekly online modules, each containing educational text, illustrative graphics, interactive exercises, and brief videos adapted from cognitive behavioural therapy for insomnia (CBT-I).
  Interventions: Behavioral: iDream2Heal
- First stage intervention: Easy Exercise (Active Comparator): Easy Exercise (eEX) is an unsupervised, self-guided web-based exercise intervention, as an active control. Through five weekly online modules, the key goals of the eEX intervention are to introduce basic sleep hygiene principals, explain the health benefit of exercise in good sleep, introduce varying levels of home-based aerobic exercise and weight training, develop a weekly exercise plan.
  Interventions: Behavioral: Easy Exercise
- Second stage intervention: Dream2Heal (Experimental): Dream2Heal (D2H) is a manualised, multi-component intervention which is grounded with core CBT-I elements of stimulus control, sleep restriction, sleep hygiene, relaxation training, and cognitive restructuring. The associations of these components with sleep improvement have been well-established in cancer population. An additional component of symptom management is incorporated, considering its co-occurrence with others physical symptoms. It consists of 5-6 weekly face-to-face sessions (45-60 min each), conducted by a trained counsellor or psychologist.
  Interventions: Behavioral: Dream2Heal
- Second stage intervention: iDream2Heal & Easy Exercise (Active Comparator): The augmented iDream2Heal & Easy Exercise (iD2H & eEX) intervention is a combined, unsupervised, self-guided web-based intervention that covers the content of iD2H and eEX interventions. It consists of the addition of an inactive intervention to a partially active intervention.
  Interventions: Behavioral: iDream2Heal & Easy Exercise

INTERVENTIONS:
Behavioral: iDream2Heal — iDream2Heal (iD2H) is an unsupervised, self-guided web-based version of the cognitive behavioural therapy for insomnia (CBT-I).
  Arms: First stage intervention: iDream2Heal
Behavioral: Easy Exercise — Easy Exercise (eEX) is an unsupervised, self-guided web-based exercise intervention.
  Arms: First stage intervention: Easy Exercise
Behavioral: Dream2Heal — Dream2Heal (D2H) is a manualised, multi-component intervention which is grounded with core CBT-I elements of stimulus control, sleep restriction, sleep hygiene, relaxation training, and cognitive restructuring.
  Arms: Second stage intervention: Dream2Heal
Behavioral: iDream2Heal & Easy Exercise — The augmented iDream2Heal & Easy Exercise (iD2H & eEX) intervention is a combined, unsupervised, self-guided web-based intervention that covers the content of iD2H and eEX interventions.
  Arms: Second stage intervention: iDream2Heal & Easy Exercise

SUMMARY:
The primary objective of this feasibility study is to assess the feasibility and acceptability, and potential clinical significance of an adaptive stepped-care intervention for improving sleep quality among Chinese cancer patients with mild-to-moderate sleep disturbance, using a sequential multiple assessment randomized controlled trial (SMART) design.

DETAILED DESCRIPTION:
The primary objective of this feasibility study is to assess the feasibility and acceptability, and potential clinical significance of an adaptive stepped-care intervention for improving sleep quality among Chinese cancer patients with mild-to-moderate sleep disturbance, using a sequential multiple assessment randomized controlled trial (SMART) design. First, the investigators will test the effect of a low intensity web-based cognitive behavioural therapy for insomnia (CBT-I) intervention (iDream2Heal; iD2H), in comparison to a low intensity web-based exercise intervention (Easy Exercise; eEX). Secondly, this study aims to explore if a stepped-up face to face, therapist led CBT-I intervention (D2H) is more effective for patients who continue to have sleep disturbance, in comparison to an augmented intervention, in which is a combined, web-based intervention that covers the content of both iD2H and eEX interventions.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese- or Mandarin-speaking Chinese patients diagnosed with curable breast, colorectal, or gynaecological cancer
* Completed treatment (except endocrine therapy) within two years
* Presenting with Pittsburgh Sleep Quality Index (PSQI) score of 6 to 11 indicating mild-to-moderate sleep disturbance

Exclusion Criteria:

* Diagnosis of metastatic cancer
* Current diagnosis of psychiatric disorder
* Current diagnosis of another sleep disorder,
* Have received psychological treatment specifically for sleep disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome (1.1) | baseline (T0)
  Rate of subject recruitment: number of participants consent and being randomized/number of eligible patients x 100
Feasibility outcome (1.2) | baseline (T0), 4-month post-intervention (T2) and 10-month post-intervention (T3)
  Rate of subject retention: number of participants who complete follow-up assessments at 4-month post-intervention (T2) and 10-month post-intervention (T3)/number of participants enrolled x 100
Feasibility outcome (1.3) | post-intervention (T1) and 4-month post-intervention (T2)
  Completion/adherence rate to intervention: number of participants who complete the intervention/number of being allocated to attend the intervention x 100
Feasibility outcome (2) | post-intervention (T1; 5 weeks post-baseline) and 4-month post-intervention (T2)
  Intervention satisfaction will be assessed using a tailored questionnaire asking whether different components of the intervention are useful, from a scale of 0-5, 1 being disagree, 5 being completely agree. Participants are also able to comment on whether the intervention's length, duration and frequency of sessions are suitable; as well as provide suggestions for areas for improvement.
Sleep disturbance | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  Sleep outcomes will be assessed using the 19-item Pittsburgh Sleep Quality Index (PSQI) evaluating specific features of sleep quality with the global score ranging from 0-21.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  HADS is a 14-item scale with seven items each for anxiety and depression subscales. Each item is scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 for anxiety or depression.
European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30) | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients. Most items are scored 1 to 4, with range of 3, with the exceptions of the items contributing to the global health status / QoL, which are scored 1-7 with a range of 6. All EORTC QLQ-C30 scale scores range from 0 to 100. A higher score for a functional scale represents a high / healthy level of functioning.

OTHER OUTCOMES:
Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  The DBAS consists of 16 items assessing sleep-related cognitions. The items are rated on a 10-point Likert scale from 0 to 10, indicating to what degree the participant agrees with the statement. Higher scores indicates more dysfunctional beliefs and attitudes. The total score is based on the average score of all items (0-10).
Global Physical Activity Questionnaire (GPAQ) | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  The GPAQ consists of 16 questions designed to estimate an individual's level of PA in 3 domains (work, transport and leisure time) and time spent in SB (Sedentary behaviour). Levels of total physical activity will be calculated using a specified formula and classified as High, Moderate or Low.
Pre-Sleep Arousal Scale (PSAS) | baseline; preintervention (T0), post-intervention (T1; 5 weeks post-baseline), 4-month post-intervention (T2) and 10-month post-intervention (T3).
  The Pre-Sleep Arousal Scale (PSAS) includes 16 items. There are two subscales, namely cognitive and somatic arousal. The response to each item ranges between 1 and 5, in which 1 = not at all and 5 = extremely. The total score ranges between 16 and 80.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- QMH department of surgery, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.